CLINICAL TRIAL: NCT06188221
Title: Does Adding Lidocaine to Corticosteroid Injections Reduce Pain Intensity in Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, David Ring, MD, PhD Associate Dean for Comprehensive Care, Professor of Surgery and Psychiatry, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-05-0094
Record Dates: First submitted 2019-07-08; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Hand Osteoarthritis; Trigger Finger; Carpal Tunnel Syndrome
MeSH Terms: conditions — Trigger Finger Disorder; Carpal Tunnel Syndrome | interventions — Lidocaine; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in two groups for the corticosteroid injection, one group with lidocaine and one group without lidocaine.
Who Masked: Participant, Care Provider
Masking Description: To make this a double-blind study, the medical assistant will put a piece of tape around the syringe to cover up the volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid with Lidocaine (Experimental): The group with the lidocaine will get a combined injection with a steroid and lidocaine. The dosages depend on the disease. The steroid dosage will be the same as for the group without lidocaine.
  * Trigger finger/De Quervain's tenosynovitis/Tendonitis: 20mg kenalog (0.5mL of kenalog 40mg/mL suspension) + 5mg lidocaine (0,5mL 10mg/mL lidocaine solution)
  * Carpal tunnel injections: 6mg betamethasone (1mL of betamethasone 6mg/mL suspension) + 20mg lidocaine (2mL 10mg/mL lidocaine solution)
  * CMC/Basal joint arthritis: 3mg betamethasone (0.5mL of betamethasone 6mg/mL suspension) + 5mg lidocaine (0,5mL 10mg/mL lidocaine solution)
  Interventions: Drug: Lidocaine; Drug: Corticoids
- Corticosteroid without Lidocaine (Active Comparator): The group without the lidocaine will get an injection with only steroids. The steroid dosage depends on the disease and will be the same as for the group with the lidocaine:
  * Trigger finger/De Quervain's tenosynovitis/Tendonitis: 20mg kenalog (0,5mL of kenalog 40mg/mL suspension)
  * Carpal tunnel injections: 6mg betamethasone (1mL of betamethasone 6mg/mL suspension)
  * CMC/Basal joint arthritis: 3mg betamethasone (0,5mL of betamethasone 6mg/mL suspension)
  Interventions: Drug: Corticoids

INTERVENTIONS:
Drug: Lidocaine — The group with the lidocaine will get a combined injection with a corticosteroid and lidocaine. The dosages depend on the disease.
  Arms: Corticosteroid with Lidocaine
Drug: Corticoids — The group without the lidocaine will get an injection with only corticosteroids. The corticosteroid dosage depends on the disease and will be the same as for the group with the lidocaine:

SUMMARY:
The purpose of this study was to determine whether adding Lidocaine to Corticosteroid injections reduce pain intensity in hand surgery.

DETAILED DESCRIPTION:
There is a lack of evidence about the use of lidocaine injection as an addition to steroids against pain during injections. Adding lidocaine adds to the volume of the injection, which might increase pain. It's possible that injecting cortisone without any lidocaine would be more comfortable than with lidocaine.

The aim of this randomized controlled trial is to assess the difference in pain intensity (during the injection and 4 hours later) between patients receiving a corticosteroid injection with or without lidocaine in patients with a hand condition. Secondarily, the aim of this study is to assess factors independently associated with pain intensity, satisfaction with the visit, and perceived empathy.

ELIGIBILITY:
Inclusion Criteria:

* All patients offered a steroid injection in a hand surgeon's office
* Aged 18-89 years
* English speaking patients
* Able to provide informed consent

Exclusion criteria:

* Non-English/Spanish speakers

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity during injection | During Injection
  11-point ordinal scale, with 0 for no pain at all and 10 for worst pain ever
Pain Catastrophizing Scale (PCS 4) | through study completion, an average of 6 weeks
  A 4 item questionnaire with a range of 0(no pain catastrophizing thoughts) to 16(maximum pain catastrophizing thoughts)
Patient Health Questionnaire (PHQ 2) | through study completion, an average of 6 weeks
  a 2 item questionnaire measuring depression symptoms with a range of 0(no depression symptoms
  0 to 6(maximum depression symptoms)
Pain Self-efficacy Questionnaire (PSEQ 2) | through study completion, an average of 6 weeks
  A measure of effective coping strategies with a range of 0(no coping strategy) to 12(maximum coping strategies)

SECONDARY OUTCOMES:
Pain intensity 4 hours after injection | 4 hours after injection
  11-point ordinal scale, with 0 for no pain at all and 10 for worst pain ever
Pain intensity 5 minutes after injection | 5 minutes after injection
  11-point ordinal scale, with 0 for no pain at all and 10 for worst pain ever

OTHER OUTCOMES:
Jefferson scale of patient perception of physician empathy | through study completion, an average of 6 weeks
  a 5 item questionnaire of patient's perceived empathy with a range of 5(minimum perceived empathy) to 35( maximum perceived empathy)

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — UT Health Austin
Locations (1):
- University of Texas Health Austin (UTHA), Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT06188221/Prot_SAP_000.pdf